CLINICAL TRIAL: NCT05252195
Title: Optimizing Detection and Prediction of Changes in Cognitive Function in Multiple Sclerosis
Brief Title: Optimizing Detection and Prediction of Changes in Cognitive Function in Multiple Sclerosis (MS)
Status: Active, not recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Wayne State University (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Anna Kratz, Associate Professor of Physical Medicine and Rehabilitation, University of Michigan
Other Study IDs: HUM00199732; 5R01HD102337-04 (NIH)
Record Dates: First submitted 2022-02-12; First posted 2022-02-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: Cognitive dysfunction
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants: Participants with Multiple Sclerosis who meet eligibility criteria.

SUMMARY:
The researchers will use technology-assisted ambulatory assessment techniques to examine cognitive dysfunction in people with Multiple Sclerosis (MS).

The researchers will determine if ambulatory assessments are sensitive to subtle declines in cognitive functioning. They will also explore the impact of modifiable factors, such as sleep, physical activity, mood, and somatic symptoms on cognitive function. These efforts will uncover behavioral and medical intervention methods. Finally, they will explore whether variability in cognitive functioning predicts short- and long-term changes in other patient-centered functional domains, social participation and physical functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Are able to fluently converse and read in English.
2. Multiple Sclerosis (MS) diagnosis (confirmed from neurologist, all relapsing and progressive subtypes included)
3. Ambulate either independently or with the use of a cane or walker (or similar device) for at least 50% of the time at baseline

Exclusion Criteria:

1. MS relapse within the past 30 days (may become eligible after 30 days; criteria used at T1, T2, and T3).
2. Inability to use study data collection tools (i.e., ActiGraph wrist-worn activity watch, smart phone app).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants include a diverse sample of patients with MS
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Function - Ambulatory measurement via Dot Memory Test | Baseline up to year 2
  Reported in terms of Euclidian distance/error
  Cognition Covariates may include: age, sex, disease duration, Multiple Sclerosis (MS) subtype (relapsing vs. progressive subtypes combined), personality variables, and cognitive reserve (education plus scores on test of vocabulary).
Change in Cognitive Function - Ambulatory measurement via Symbol Search Test | Baseline up to year 2
  Reported in Reaction Time (milliseconds)
  Cognition Covariates may include: age, sex, disease duration, Multiple Sclerosis (MS) subtype (relapsing vs. progressive subtypes combined), personality variables, and cognitive reserve (education plus scores on test of vocabulary).
Change in Cognitive Function - clinic-based neurocognitive measurement via NIH Toolbox Cognitive Battery | Baseline up to year 2
  Test Battery reported in T-scores. Covariates may include: age, sex, disease duration, MS subtype (relapsing vs. progressive subtypes combined), personality variables, and cognitive reserve (education plus scores on test of vocabulary).
Change in Cognitive Function - clinic-based neurocognitive measurement via Symbol Digit Modalities test | Baseline up to year 2
  Covariates may include: age, sex, disease duration, MS subtype (relapsing vs. progressive subtypes combined), personality variables, and cognitive reserve (education plus scores on test of vocabulary).
  The score is the number of correct answers in 90 seconds. Higher scores indicates better attention and processing speed.
Change in Cognitive Function - clinic-based neurocognitive measurement via Paced Auditory Serial Addition Test | Baseline up to year 2
  Covariates may include: age, sex, disease duration, MS subtype (relapsing vs. progressive subtypes combined), personality variables, and cognitive reserve (education plus scores on test of vocabulary).
  The score range is 0-60 and higher numbers indicate better sustained attention, speed of information processing, and working memory.
Change in Cognitive Function - clinic-based neurocognitive measurement via Rey Auditory Verbal Learning Test | Baseline up to year 2
  Covariates may include: age, sex, disease duration, MS subtype (relapsing vs. progressive subtypes combined), personality variables, and cognitive reserve (education plus scores on test of vocabulary).
  The scores from the test represent the total immediate recall (over 5 learning trials), delayed recall, and recognition. Higher scores indicate better verbal learning and memory.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kratz, Principal Investigator — University of Michigan; Nora Fritz, Principal Investigator — Wayne State University
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kratz AL, Ehde DM, Alschuler KN, Pickup K, Ginell K, Fritz NE. Optimizing Detection and Prediction of Cognitive Function in Multiple Sclerosis With Ambulatory Cognitive Tests: Protocol for the Longitudinal Observational CogDetect-MS Study. JMIR Res Protoc. 2024 Sep 26;13:e59876. doi: 10.2196/59876. PMID 39325510